CLINICAL TRIAL: NCT05829161
Title: Sensory Phenotypes of Autism Spectrum Disorder Across Lifespan: Prospective Cohort Study and Sensory-Social Paradigm Establishment
Brief Title: Sensory Phenotypes of Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201903126RINA
Record Dates: First submitted 2019-07-04; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD Group: ASD participants, no intervention
  Interventions: Behavioral: no intervention
- TD Group: TD participants, no intervention
  Interventions: Behavioral: no intervention

INTERVENTIONS:
Behavioral: no intervention — no intervention

SUMMARY:
This project plans to establish sensory phenotypes of a Taiwanese ASD cohort across lifespan, including variety of sensory modalities, sensory domains, and clinical correlates.

Also, we will clarify the relationship between sensory phenotypes and social impairment by two specific sensory-social paradigms targeting eye gaze avoidance and social touch anxiety, as well as the atypical neural representation of ASD during eye gaze and viewing social touch by fMRI and EEG.

DETAILED DESCRIPTION:
Sensory disturbance of autism spectrum disorder (ASD) are life-long highly-impairing challenges for the individual. Anxiety and fear around the sensory issues significantly threatens the psychological and mental health. As a newly introduced diagnostic criteria of ASD, sensory characteristics becomes a recent focus of ASD research. The ASD population is aging, how their sensory features naturally change with age is particular relevant for their adaptation. However, current literature are limited to childhood and young adults and mostly rely on behavioral report, lacking a clear whole picture of changing sensory phenotype in terms of different sensory modality and sensory domains. Besides, how sensory characteristics in ASD can be quantified by objective measures or explored by qualitative approach, how the sensory sensitivity contributes to the core social deficits in ASD such as eye gaze or social touch avoidance are unclear. This project plans to achieve the following aims:

1. Establish sensory phenotypes of a Taiwanese ASD cohort across lifespan, including variety of sensory modalities (i.e., visual, tactile, auditory, smell/taste, proprioception, etc.), sensory domains (i.e., low registration, sensory seeking, sensory sensitivity, and sensory avoiding), and clinical correlates.
2. Clarify the relationship between sensory phenotypes and social impairment by two specific sensory-social paradigms targeting eye gaze avoidance and social touch anxiety, which are hallmarks of ASD. Factors of emotion types as well as familiarity of faces or social/object touch will be manipulated to examine how they moderate eye tracking and pupil response.
3. Identify the atypical neural representation of ASD during eye gaze and viewing social touch by fMRI and EEG.

ELIGIBILITY:
Aim#1

Inclusion Criteria:

* Diagnosis of autism spectrum disorder Aim#2 and #3

ASD group:

Inclusion Criteria:

* Diagnosis of autism spectrum disorder
* Age above 12-40 years old

Exclusion Criteria:

* No diagnosis of autism spectrum disorder
* Pregnant woman
* Metal implant in the body

TD group:

Inclusion Criteria:

* No diagnosis of autism spectrum disorder
* Age above 12-40 years old

Exclusion Criteria:

* History of major psychiatric disorders
* Pregnant woman
* Metal implant in the body

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with autism spectrum disorder, recruited from National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-07-12 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile | 2 years
  It is a self-report scale covers 6 sensory modalities, including taste/smell, motion, visual, tactile, activity, and auditory sensation. The scoring method was based on 4-dimension structure, i.e. Low Registration, Sensation Seeking, Sensory Sensitivity, and Sensation Avoiding. Higher scores mean worse symptoms for each dimension compared to average healthy controls

SECONDARY OUTCOMES:
Brain activation through fMRI data | 2 years
  MRI scanning session consist of eye-avoidance paradign, social touch paradigm and anatomical scan. Regions of interest for eye avoidance paradigm included brain regions that have been shown to involve face-to-face social and emotional interaction. ROIs for social touch paradigm select the areas that are known to mediate the processing of visually presented social touch scenes.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ling Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan